CLINICAL TRIAL: NCT03032484
Title: A Phase 2 Investigator Initiated Study to Determine the Efficacy and Safety of TVB- 2640 in Combination With Bevacizumab in Patients With First Relapse of High Grade Astrocytoma
Brief Title: TVB- 2640 in Combination With Bevacizumab in Patients With First Relapse of High Grade Astrocytoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 16-0136
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Astrocytoma
MeSH Terms: conditions — Astrocytoma | interventions — Bevacizumab; TVB-2640

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bevacizumab and TVB-2640 (Experimental): Bevacizumab every 2 weeks in combination with TVB-2640 dosed at 100mg/m2 daily (rounded to 50mg tab dose), from day 1 until day 28 of the first cycle.
  Interventions: Drug: Bevacizumab; Drug: TVB-2640
- Bevacizumab for Cycle 1, then Bevacizumab and TVB-2640 (Experimental): Bevacizumab alone every 2 weeks, on days 1 and 15 until day 28 of the first cycle, and then receive both Bevacizumab and TVB-2640 for the remainder of their participation in this study.
  Interventions: Drug: Bevacizumab; Drug: TVB-2640

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab is FDA approved as a treatment for recurrent Glioblastoma following failure of radiation therapy and temozolomide.
  Other Names: Avastin
Drug: TVB-2640 — TVB-2640 is a potent and reversible inhibitor of the FASN enzyme. TVB-2640 inhibits the β-ketoacyl reductase (KR) enzymatic activity of the FASN enzyme.

SUMMARY:
Randomized phase 2 study TVB-2640 in combination with Bevacizumab versus Bevacizumab alone.

DETAILED DESCRIPTION:
Eligible patients will be randomized into 2 separate arms:

* Arm number one will receive Bevacizumab every 2 weeks in combination with TVB-2640 from day 1 until day 28 of the first cycle.
* Arm number two will receive Bevacizumab alone every 2 weeks, from on days 1 and 15 of the first until day 28 of the first cycle.
* MR-Spectroscopy will be obtained on all patients (both arms) at day 28 of first cycle.
* Starting on cycle 2 day 1, all patients will converge to a single arm and will continue to receive bevacizumab every 2 weeks in combination with TVB-2640. Every cycle will last 28 days.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee
* Histologically confirmed high-grade astrocytoma
* Progression following standard combined modality treatment with radiation and temozolomide chemotherapy
* Recovered from reversible toxicities of prior therapy to Grade 0 or Grade 1
* ECOG Performance Status of 0 to 2
* Life expectancy of at least 3 months
* Adequate renal and liver function: AST/ALT ≤ 3 x ULN, Bilirubin ≤ 1.5 times ULN, Creatinine ≤ ULN
* Adequate hematologic status (without hematologic support): Hemoglobin ≥ 9 g/dL, ANC ≥ 1500 cells/ml, Platelets ≥ 100,000 cells/ml
* All women of childbearing potential must have a negative serum pregnancy test and male and female subjects must agree to use effective means of contraception (for example, surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through six months after the last dose.

Exclusion Criteria:

* Receiving warfarin (or other coumarin derivatives) and is unable to switch to low molecular weight heparin (LMWH) before the first dose of study drug
* Evidence of acute intracranial or intratumoral hemorrhage either by MRI or CT scan. Subjects with resolving hemorrhage changes punctuate hemorrhage, or hemosiderin are eligible
* Unable to undergo MRI scan (e.g., pacemaker)
* Received enzyme-inducing anti-epileptic agents within 14 days of study drug (e.g., carbamazepine, phenytoin, phenobarbital, primidone)
* Not recovered to a NCI CTCAE v.4.03 Grade ≤ 1 from AEs (except alopecia and lymphopenia) due to surgery, antineoplastic agents, investigational drugs, or other medications that were administered prior to study drug
* Evidence of wound dehiscence
* Pregnant or breast-feeding
* Clinically significant Dry Eye or necessary contact lens use
* Serious intercurrent illness such as: Hypertension (two or more blood pressure readings performed at screening of > 150 mmHg systolic or > 100 mmHg diastolic) despite optimal treatment, Non-healing wound or ulcer, Uncontrolled life threatening cardiac arrhythmias, Untreated hypothyroidism, Uncontrolled active infection, Symptomatic congestive heart failure or unstable angina pectoris within 3 months prior to study drug, Gastrointestinal perforation, abdominal fistula, intra-abdominal abscess within 1 year
* Inherited bleeding diathesis or coagulopathy with the risk of bleeding
* HIV , Hepatitis B or C documented infections
* Received any of the following prior anticancer therapy: Non-standard radiation therapy such as brachytherapy, systemic radioisotope therapy (RIT), or intra-operative radiotherapy (IORT). Note: stereotactic radiosurgery (SRS) is allowed, Non-antiangiogenic therapy (including investigational agents and small molecular kinase inhibitors) within 7 days or 5 half-lives, whichever is shorter, prior to the first dose of study drug, Biologic agents (antibodies, immune modulators, vaccines, cytokines) within 21 days prior to first dose of study drug, Nitrosoureas or mitomycin C within 42 days or metronomic/protracted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2020-04-04 (Actual); Study Completion 2021-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Brenner, Principal Investigator — UT Health San Antonio
Locations (1):
- University of Texas Health Science Center San Antonio at the Cancer Therapy and Research Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A cycle 1 randomization to either TVB-2640 plus bevacizumab or bevacizumab monotherapy was conducted in this trial. This randomization was performed for biomarker analysis only and was not intended to be comparative for either safety or efficacy, as it would be unexpected to observe a difference in survival after only one cycle of a study drug.
Groups:
- Bevacizumab: Bevacizumab alone every 2 weeks, on days 1 and 15 until day 28 of the first cycle.
  Bevacizumab: Bevacizumab is FDA approved as a treatment for recurrent Glioblastoma following failure of radiation therapy and temozolomide.
Period: Overall Study Cycle 1 (C1)
Arm/Group | Bevacizumab and TVB-2640 | Bevacizumab
Started (After C1, all subjects were treated with a combination of TVB-2640 with Bevacizumab) | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Start of Second Cycle (C2)
Arm/Group | Bevacizumab and TVB-2640 | Bevacizumab
Started (All subjects were aggregated from Arms 1 and 2 into a single treatment group from cycle 2 onwards, and efficacy and safety data were assessed for the aggregated group.) | 24 (All subjects were treated with TVB-2640 and Bevacizumab following C1, there was no continuation of Bevacizumab treatment alone, and efficacy and safety data were assessed for the aggregated group.) | 0 (All subjects were treated with TVB-2640 and Bevacizumab following C1. No subject progressed to Bevacizumab treatment alone, all were treated with TVB/Bev combination.)
Completed | 23 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab and TVB-2640
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 61 [37 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival at 6 Months (PFS6)
Description: Survival of participants at 6 months after the start of treatment without their condition becoming any worse. Brain magnetic resonance imaging (MRI) was performed after every even cycle (e.g., C2, C4) during treatment, with tumor response assessed by the investigator for complete response (CR), partial response (PR) and PD according to the Response Assessment in Neuro-oncology (RANO) criteria.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab and TVB-2640
Number analyzed (Participants) | 23
percentage of participants | 47

2. Secondary Outcome: Incidence, Nature and Severity of Adverse Events and Serious Adverse Events, Graded According to NCI - Common Toxicity Criteria for Adverse Events Version (4.03)
Description: Number of adverse of any nature are reported as well as the number of adverse events that were classed as grade 3-5 on the NCI - Common Toxicity Criteria for Adverse Events
Time Frame: Up to 6 28-day cycles
Population: Subject who received TVB-2640 and Bevacizumab or Bevacizumab alone
Measure: Number; unit: number of events
Arm/Group | Bevacizumab and TVB-2640
Number analyzed (Participants) | 23
number of events
  Number of adverse events any grade | 183
  Adverse events grade 3-5 | 27

3. Other Pre Specified Outcome: Metabolic Change Analysis of Tumor Tissue by MRS (Magnetic Resonance Spectroscopy)
Description: The MRI was performed during cycle 2. This procedure was intended to be outsourced, and MRIs performed locally produced inadequate resolution, so no data analysis was obtained from this measure.
Time Frame: Cycle 2: approximately 56 days
Population: Data were not evaluable for this measure, since MRI resolution was inadequate
Arm/Group | Bevacizumab and TVB-2640
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study enrollment for up to six cycles (28 days each) or until there is evidence of significant treatment related toxicity or progressive disease. Subject were assessed for adverse events which occurred after the start of treatment until 30 days after study drug discontinuation or subsequent cancer therapy was initiated. Adverse events were collected over a 1.5 year period.
Description: Bevacizumab during cycle 1 and Bevacizumab and TVB-2640 were combined as pre-specified in the study protocol
Arm/Group | Bevacizumab and TVB-2640
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 4/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and TVB-2640 (N=23)
Aphasia (Nervous system disorders) | 1 (1)
Thromboembolic event (Blood and lymphatic system disorders) | 1 (1) — Right lower extremity deep vein thrombosis
Vomiting (Gastrointestinal disorders) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) — Perirectal abcess
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab and TVB-2640 (N=23)
Palmar plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 18 (41)
Mucositis (Skin and subcutaneous tissue disorders) | 15 (22)
Hypertension (Cardiac disorders) | 13 (21)
Dry Eye (Eye disorders) | 12 (13)
Fatigue (General disorders) | 7 (9)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Skin infection (Skin and subcutaneous tissue disorders) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Elevated ALT/AST (Hepatobiliary disorders) | 3 (3) — Elevated liver enzymes
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (3)
Depression (Nervous system disorders) | 3 (3)
Dysphasia (Gastrointestinal disorders) | 3 (3)
Headache (General disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Parestheisa (Musculoskeletal and connective tissue disorders) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 2 (4)
Cognitive Disturbance (Nervous system disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 2 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Limb edema (Blood and lymphatic system disorders) | 2 (2)
Hypokalemia (Renal and urinary disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Increased Creatinine (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT03032484/Prot_SAP_000.pdf